CLINICAL TRIAL: NCT00318864
Title: Stress, the HPA and Health in Aging
Brief Title: Biological CVD Risk Factors in Older Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CBarrTaylor; 5P01AG018784-02 (NIH)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Depression; Hypertension; Hypercholesterolemia
Keywords: depression; cardiovascular risk; mechanisms
MeSH Terms: conditions — Depression; Hypertension; Hypercholesterolemia | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy

SUMMARY:
The purpose of this study is to determine if improvements in mood will ameliorate autonomic dysregulation, HPA dysfunction and typical (e.g. lipids) and atypical risk factors in depressed patients with elevated cardiovascular risk (CVD). Up to 70, depressed participants with elevated cardiovascular risk factors were randomized to a cognitive behavioral intervention (CBT) or a waiting list control (WLC) condition. Twenty non-depressed age and risk-matched controls will also recruited. Traditional risk factors (e.g. lipids, blood pressure, heart rate), atypical risk factors (endothelial function, asymmetric dimethylarginine, C-reactive protein) will be measured pre and post treatment six months later Subjects will undergo a psychophysiological stress test while cardiovascular physiology was measured. Salivary cortisol will be measured during the day and during the psychological stress test. Depressed subjects will be randomized to a 16 week cognitive behavior therapy intervention or to a wait-list control. It is hypothesized that reduction in mood will be associated with reduction in typical and atypical risk factors.

DETAILED DESCRIPTION:
Recruitment:

The sample will be drawn from the following Stanford Health Services clinics: the Stanford Cardiovascular Risk Reduction Clinic, the Electron Beam Computed Tomography Center, and the Cardiology Clinics. Subjects will also be recruited via the mass media.

Screen:

Potential subjects will be identified by a brief screen combined with a short follow-up interview, the PRIME-MD that consists of two self-report items, as follows: "During the PAST MONTH, have you been bothered A LOT by (1) little interest or pleasure in doing things (yes or no) or (2) feeling down, depressed, or hopeless (yes or no)." If either item is scored "yes," a short follow-up interview to establish a diagnosis is indicated. The two screen items yield a sensitivity of 69% and specificity of 82% when diagnoses made by a mental health professional are used as the criterion standard. Subjects will also have to have a general health questionnaire score > 5, indicating high levels of distress. Potentially eligible subjects will then undergo a structured clinical interview for diagnosis. Twenty, age, gender and cardiovascular risk level controls will be selected from the same population. Controls will be matched for age, sex and risk with the depressed subjects.

Procedures:

Participants will come to the Department of Psychiatry for baseline assessment, including undergoing a structured psychiatric examination and completing baseline self-report measures. If they are interested and eligible they will be asked to complete a series of assessments that will last three days. On day one, they will then be asked to report to the Stanford General Research Center on their next available Wednesday, at 9:00. At that time a medical exam will be performed, bloods were will be drawn and the FMVD (see below) undertaken. They will then be asked to wear a the "lifeshirt," a undergarment worn over the chest that will measure heart rate during the day, and to report their mood and activity on up to 5 occassions using a portable computer attached to the lifeshirt. Each participant will be scheduled to obtain saliva samples using cotton swabs in "salivette devices" at the time of waking, 30 minutes later, and then at 1200h, 1700h, and 2100h on each of two days. Participants were asked to refrigerate each sample immediately after collection, not to eat, drink, smoke, brush their teeth, or use mouthwash in the 30 minutes before collection, and not to drink alcohol during the 8-10 hours prior to collecting samples or during the days of collection. On day two they will return the life-shirt and continue to obtain salivary cortisols. On day three they will be asked to return to the Stanford GCRC to undertaken a psychological stress test. The psychological stress test is a standardized social and cognitive stressor composed of 5 minutes of anticipatory stress, and then 5 minutes of public speaking (simulated job interview) and 5 minutes of mental arithmetic, both done before a panel of 2 evaluators. Subjects were sitting in a comfortable chair throughout the entire procedure. Subjects were informed that their speech would be evaluated by a panel of two expert behavioral coders and that it would be rated on the basis of poise, speaking ability, and expressiveness. During the psychological stress a number of physiologic functions will be measured using sensors attached to the chest and arms. Subjects will also be asked to provide saliva samples between the measurements and to report their mood. At the end of the stress testing they will meet with an investigator to be debriefed.

Depressed subjects randomized to the cognitive behavior therapy (CBT)will be asked to attend 16, one-hour sessions over 4-5 months. The CBT will be conduced by a senior therapist. Cognitive therapy aims at symptom removal by identification and correction of the patient's distorted, negatively biased, moment-to-moment thinking and theoretically aims at prevention of relapse/reoccurrence by identifying and correcting silent assumptions (personal beliefs or schemas). Modern cognitive treatment interventions also address behavioral aspects of depression through encouraging more activity of various kinds. (Because the level of physical condition is a potential confound for the variables of interest, increased aerobic activity will not be included in the intervention.) Depressed control subjects will be offered the CBT intervention (in a group format) after the six-month follow-up and/or referred for treatment, as desired and appropriate. At post-treatment and six-month follow-up, subjects will be carefully assessed for any psychotherapy and psychopharmacology interventions.

The same assessments will be conducted at baseline and six months later.

Measures:

Intervention Descriptive and Control Variables: Baseline demographic information will include education, ethnicity and marital status.

Structured Clinical Interview for Diagnosis (SCID). A structured clinical interview for diagnosis modified to include the Hamilton Depression Interview will be used. Structured clinical interviews are now the standard method of diagnosis in psychiatry studies.

Medical status. A standard questionnaire concerning coronary risk factors, medications, and medical diagnosis will be completed at baseline on all subjects. Heart rate and baseline ECG. Resting 12-lead ECG will be recorded using a standard electrocardiograph at the time of the treadmill. Subjects with CVD events evident on their ECG will be excluded. Blood pressure. Resting blood pressure will be measured in triplicate by asculatory techniques using a mercury sphygmomanometer.

Body weight (kg) and height (m). Weight (in kgs) will be measured on a balance beam scale. Height and weight will be obtained in a standing position, with shoes removed and subjects wearing street clothes.

Lipids and apolipoproteins. Fasting plasma levels of total cholesterol and triglycerides will be obtained from fasting samples.

Duplex ultrasonography of flow-mediated vasodilation (FMVD). The methods are as follows: Diameter of the brachial arterial (DBA) will be measured at multiple single time points under 4 states using a standard 7 MHz linear array transducer and a Hewlett-Packard system (Hewlett-Packard, Palo Alto, California). The four states include: at rest, during limb ischemia (created by inflating a blood pressure cuff placed distal to the brachial artery to supra-systemic pressures), in response to reactive hyperemia (with increased flow producing endothelium-dependent vasodilation). Measurements of these three states will then be repeated a second time. Finally, DBA will then be measured in (4) response to the administration of sublingual nitroglycerin. ADMA (asymmetric dimethylarginine) will be measured.

Hypothalamic-Pituitary-Adrenal Axis Activity Cortisol and diurnal cortisol variation. Cortisol will be measured using self-administered saliva samples. Subjects will obtain samples on three consecutive days, at five intervals throughout each day (at waking, 45 minutes later, 5 pm, 9 pm and bedtime), in subjects' own homes. A testing kit will be used by each subject consisting of 15 salivette tubes. Salivary cortisol has been found to be a reliable tool for investigations of hypothalamic-pituitary-adrenal axis activity.

Laboratory Assessment of RSA and Baroreflex Sensitivity RSA and baroreflex sensitivity will be assessed noninvasively in the laboratory during a 10-minute baseline. Physiological channels required for their quantification will be recorded using (1) an ECG (400 Hz sample rate); (2) two channels of respiration using a Respitrace system (Ambulatory Monitoring, Ardsley, NY); bands are placed around the upper thorax and around the abdomen and calibrated against spirometry (25 Hz sample rate); (3) a continuous arterial blood pressure waveform from the index finger by means of the Finapres 2300 system.

Depression measures include the Hamilton Depression Interview (HDI) and the Beck Depression Interview (BDI), a short 21-item will also be obrtained. Perceived Stress Perceived Stress Scale (PSS). The PSS measures a global perception of stress during the previous month. It has a short version comprised of ten items, e.g., "In the last month how often have you felt difficulties were piling up so high that you could not overcome them?" Response options were assessed using a 5-point Likert-type scale: (0 = Never to 4= Very Often). The scores on four items that were worded in the opposite direction (e.g., "In the last month how often have you felt that things were going your way?") are reverse-scored.

ELIGIBILITY:
Inclusion Criteria:

* age > 55 years, hypertensive or hypercholesterolemic, depressed

Exclusion Criteria:

* suicidal

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-06; Study Completion 2005-07

PRIMARY OUTCOMES:
Change in depression

SECONDARY OUTCOMES:
Change in typical and atypical risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Craig B Taylor, Principal Investigator — Stanford Medical Center
Locations (1):
- Stanford Medical Center, Stanford, California, United States